CLINICAL TRIAL: NCT04935931
Title: Eating Disorder Individualized Therapeutics-Naltrexone Neuroimaging (EDIT-N2)
Brief Title: Naltrexone Neuroimaging
Acronym: EDIT-N2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Stephani Stancil, Assistant Professor, Children's Mercy Hospital Kansas City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00001668; UL1TR002366 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Eating Disorders; Binge Eating; Purging (Eating Disorders)
Keywords: Pediatric; Adolescent; Eating Disorder; Neuroimaging; Naltrexone
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot (Experimental): Pre/post fMRI
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — naltrexone 50 mg PO x 1

SUMMARY:
The purpose of this open-label, pilot study is to evaluate fMRI as a biomarker of opioid antagonism in adolescents with ED. Modulation of brain activation will be examined in regions of interest by fMRI using a food-specific and general reward task in adolescents with ED in a pre/post design.

DETAILED DESCRIPTION:
This is an open-label, interventional trial to evaluate reward system modulation (detected by neuroimaging) in response to opioid antagonism (i.e., naltrexone) in adolescents aged 13-21 years with an eating disorder characterized by the target behaviors of binge eating and/or purging (e.g., AN-BP, BN, BED). A pre/post design completed on the same day will be employed to quantify within-individual change while reducing potential confounding due to known neuroimaging variables (e.g., menstrual phase, treatment changes) that may occur with time elapsed between study visits. Self-report data regarding will be captured via electronic surveys using validated instruments (where possible), structured interview, study records.

Reward System Modulation by fMRI. Each scan will last approximately 1 hour and involve two reward activation paradigms: passive food view (PFV) and monetary incentive delay (MID). These two reward activation paradigms provide distinct insight and will generate pilot data to support the choice of the optimal paradigm for further testing of reward system modulation in adolescents with eating disorders. PFV provides a paradigm that is relevant to the target behaviors (i.e., binge eating, purging), has been evaluated in ED patients, in response to naltrexone in adults, and is expected to activate food cue-reactivity regions (e.g., prefrontal cortex). MID is a widely used paradigm in adolescents to detect reward anticipation and receipt particularly in the striatum and is currently being used to study the developmental trajectory of reward processing in the longitudinal Adolescent Brain Cognitive Development (ABCD) trial. To the greatest extent possible, we will harmonize our fMRI parameters with those published for ABCD.

Opioid Antagonism and exposure-response linkage. A single oral dose of naltrexone hydrochloride 50 mg tablet will be administered. Plasma and urine will be obtained to measure systemic exposure to naltrexone and it primary, active metabolite, 6-beta-naltrexol, using a validated UPLC-MS/MS assay.

ELIGIBILITY:
Inclusion Criteria:

* Eating disorder diagnosis per DSM-V criteria that is characterized by binge eating (defined as loss of control of eating resulting in large amount of food consumed in a short period of time) and/or purging (e.g., vomiting, excessive exercising, laxative use)
* Stable medication regimen (no dose or drug changes in the past 4 weeks)
* Participant and parent/legal guardian (if under 18 years) are willing and able to provide informed permission/assent/consent for the study

Exclusion Criteria:

* Pregnant (via UCG)
* Prior hypersensitivity reaction to naltrexone (e.g., anaphylaxis)
* Non-removable metal in the body
* Current naltrexone use
* Self-reported opioid use in the past 7 days
* A language barrier (e.g., non-English speaking) for the participant that precludes communication and/or ability to complete all study-related requirements.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephani Stancil, PhD, Principal Investigator — Children's Mercy Kansas City
Locations (1):
- Children's Mercy Research Institute, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Stancil SL, Yeh HW, Brucks MG, Bruce AS, Voss M, Abdel-Rahman S, Brooks WM, Martin LE. Potential biomarker of brain response to opioid antagonism in adolescents with eating disorders: a pilot study. Front Psychiatry. 2023 Jul 10;14:1161032. doi: 10.3389/fpsyt.2023.1161032. eCollection 2023. PMID 37492067

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Pre/Post Design: Pre-naltrexone fMRI
  Naltrexone: naltrexone 50 mg PO x 1
  Post-naltrexone fMRI
Period: Overall Study
Arm/Group | Single Pre/Post Design
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Pre/Post Design
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (2.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender identity: Female | 12
  Gender identity: Male | 0
  Gender identity: Other (prefer to self-describe) | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in % Blood Oxygenation Level Dependent Change (%BOLD) in the Nucleus Accumbens
Description: Change in %BOLD following single dose naltrexone (post-pre) within individuals during passive food view task in the nucleus accumbens
Time Frame: 2 hours post-naltrexone vs baseline
Measure: Mean (Standard Deviation); unit: %BOLD signal change
Arm/Group | Single Pre/Post Design
Number analyzed (Participants) | 12
%BOLD signal change | -0.08 (0.03)

2. Primary Outcome: Change in % Blood Oxygenation Level Dependent Change (%BOLD) in the Dorsal Anterior Cingulate Cortex
Description: Change in %BOLD following single dose naltrexone (post-pre) within individuals during monetary incentive delay in dorsal anterior cingulate cortex
Time Frame: 2 hours post-naltrexone vs baseline
Measure: Mean (Standard Deviation); unit: %BOLD signal change
Arm/Group | Single Pre/Post Design
Number analyzed (Participants) | 12
%BOLD signal change | 0.06 (0.03)

3. Secondary Outcome: Exposure
Description: Maximum plasma concentration of naltrexone at 2 hours post-single dose
Time Frame: 2 hours post-naltrexone
Population: plasma concentration
Measure: Mean (Standard Deviation); unit: nanomolar
Groups:
- Single Pre/Post Design: Naltrexone 50 mg PO x 1, blood collected 2 hours post-dose
Arm/Group | Single Pre/Post Design
Number analyzed (Participants) | 12
nanomolar | 44.1 (22.7)

ADVERSE EVENTS:
Time Frame: 1 day (single study visit)
Arm/Group | Single Pre/Post Design
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Pre/Post Design (N=13)
Claustrophobia (Nervous system disorders) | 1 (1) — Claustrophobia during MRI

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/31/NCT04935931/Prot_SAP_ICF_000.pdf